CLINICAL TRIAL: NCT04929132
Title: Added Value of Contrast-enhanced Ultrasound for BI RADS 4A Nodules Graded With the Breast Imaging Reporting and Data System
Brief Title: Added Value of Contrast-enhanced Ultrasound for BI RADS 4A Nodules
Acronym: BIRADS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHZhejiangU 123
Record Dates: First submitted 2021-04-07; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-12

CONDITIONS: Ultrasound; Breast Cancer; Pathology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — pathology results of breast nodules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to investigate the added value of contrast-enhanced ultrasound (CEUS) for differentiating low risk patients with breast nodules categorized as 4A using the Breast Imaging Reporting and Data System (BI-RADS).

DETAILED DESCRIPTION:
The aim of this study was to investigate the added value of contrast-enhanced ultrasound (CEUS) for differentiating low risk patients with breast nodules categorized as 4A using the Breast Imaging Reporting and Data System (BI-RADS). The study included patients with 4A nodules confirmed by core biopsy and/or surgery. The CEUS parameters were assessed to evaluated the added value in BI-RADS 4A nodules

ELIGIBILITY:
Inclusion Criteria:

patients with nodules which were sonographically classified as BI-RADS 4 A breast lesion

Exclusion Criteria:

(i) absence of a pathologic diagnosis; (ii) presence of breast nodules that were too large to compare with normal parenchyma; (iii) patients with radiotherapy and chemotherapy of breast cancer; and (iv) skin disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with nodules which were sonographically classified as BI-RADS 4 A breast lesion
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
CEUS | up to 3 months
  if the result of CEUS is positive，the nodule was downgraded. if the result of CEUS is negative, the nodule was kept as BI RADS 4A category. Then all nodules were submitted to biopsy or surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZJU, Hanzhou, Zhejiang, China